CLINICAL TRIAL: NCT06313346
Title: Effect of a Probiotic Consumption on Microbiota Associated with the Immune System and Inflammation in Adult Women and Men (FLORABIOTIC INMUNITARIO).
Brief Title: Effect of a Probiotic on Microbiota Associated with the Immune System and Inflammation.
Acronym: FLORABIOTIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2023.200
Record Dates: First submitted 2024-03-01; First posted 2024-03-15 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2023-12

CONDITIONS: Probiotic; Microbiota
Keywords: Microbiota; Probiotic; Inflammation; Immune system; Humans; Randomized controlled trial; Cortisol
MeSH Terms: conditions — Inflammation | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Randomised, double blinded, parallel intervention
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The products (experimental and placebo), will be produced by an external producer, who will save the codes. None of the researchers involved in the study development or analyses will know the association until the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic group (Experimental): Subjects will consume one capsule of probiotic, daily, during 6 weeks.
  Interventions: Dietary Supplement: Probiotic
- Placebo group (Placebo Comparator): Subjects will consume one capsule of placebo, daily, during 6 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Probiotic capsules
  Arms: Probiotic group
Dietary Supplement: Placebo — Placebo capsules
  Arms: Placebo group

SUMMARY:
The goal of this randomized clinical trial is to learn about the effect of consuming a probiotic on the microbiota associated with immune health and inflammation in healthy women and men after 6 weeks of intervention.

The main questions to answer are:

1. To study changes in the intestinal microbiota associated with immune health and inflammation related to probiotic intake.
2. To evaluate changes in salivary cortisol after ingestion of the probiotic.
3. To compile the number and intensity of catarrhal episodes suffered by the participants along the study.

For this purpose, a randomized, double blind parallel study has been designed.

Target sample size is 60 subjects.

Participants will be allocated in two groups for 6 weeks:

* Experimental group (n=30): daily consumption of one probiotic capsule.
* Placebo group (n=30): daily consumption of one placebo capsule.

DETAILED DESCRIPTION:
Volunteers who wish to participate in the study will be interviewed by phone to verify that they meet the main inclusion criteria. Volunteers who meet the main inclusion criteria will be invited to an information and screening visit to resolve any doubts. Volunteers who agree to participate in the study will sign the informed consent and will be randomly allocated to one of the two arms of the study and will be provided with any required material.

During the intervention, volunteers will attend two Clinical investigation visits. The first one will be carried out on the first day of the study and the last one will take place at the end of the 6 weeks. In both visits anthropometric and body composition measurements, stool and saliva samples, as well as data about dietary, physical activity and catarrhal episodes will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers of both sexes.
* Age between 40 and 65 years old.
* Volunteers with a body mass index between 18.5 and 30 kg/m2.
* Subjects have to present a stable weight (+/- 3 kg) in the last three months prior to the start of the study.
* Subjects must be able to understand and be willing to sign the informed consent, and comply with all study procedures and requirements.

Exclusion Criteria:

* Subjects with relevant functional or structural anomalies of the digestive system, such as malformations, angiodysplasias, active peptic ulcers, chronic inflammatory or malabsorption diseases, hiatal hernia, reflux, etc.
* Subjects with surgical interventions with permanent consequences in the digestive system (for example, gastroduodenostomy).
* Subjects following treatments that alter gastrointestinal function, either chronically or occasionally.
* Subjects who are being treated with antibiotics (in order to participate, they do not have to have taken antibiotics during the two months prior to the baseline visit).
* Subjects with any type of cancer or undergoing treatment for it, or less than 5 years since its eradication.
* Subjects with any liver disease (may participate with non-alcoholic fatty liver disease).
* Subjects with allergy to any component of the product under study.
* Subjects with a high alcohol intake, more than 14 units (women)/day and 20 units (men)/day.
* Women who are breastfeeding or pregnant.
* Subjects who present some type of cognitive and/or psychological impairment.
* Subjects with poor collaboration or with difficulties for following the study procedures.
* Subjects who work with shift changes that include nights.
* Subjects who follow any type of supplementation that interferes with the study (example: consumption of probiotics).
* Subjects who are immersed in diet/exercise changes.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Fecal microbiota | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Fecal microbiota of participants will be analyzed by bacterial 16S gene sequencing technology.

SECONDARY OUTCOMES:
Salivary cortisol | Clinical Investigation Day 1 (at wake up in the morning) and Clinical Investigation Day 2 (at wake up in the morning, at the same time taken in the clinical investigation day 1)]
  Cortisol levels will be taken by Salivette®- Cortisol kit and analyzed by electrochemiluminescence immunoassay and reported in ug/dL.
Body weight | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Weight of participants will be measured by bioimpedance and reported in kg
Height | Clinical Investigation Day 1.
  Height of participants will be measured by stadiometer and reported in m.
Body mass index | Clinical Investigation Day 1 and Clinical Investigation Day 2.
  Body mass index will be calculated as follows: weight (kilograms)/ height (cm)2.
Body fat percentage | Clinical Investigation Day 1 and Clinical Investigation Day 2.
  Body fat of participants will be analyzed by bioimpedance and reported in percentage and kilograms.
Body muscle mass | Clinical Investigation Day 1 and Clinical Investigation Day 2.
  Body muscle mass of participants will be analyzed by bioimpedance and reported in kilograms.
Body lean mass | Clinical Investigation Day 1 and Clinical Investigation Day 2.
  Body leen mass of participants will be analyzed by bioimpedance and reported in kilograms.
Body water mass | Clinical Investigation Day 1 and Clinical Investigation Day 2.
  Body water mass of participants will be analyzed by bioimpedance and reported in kilograms.
Body bone mass | Clinical Investigation Day 1 and Clinical Investigation Day 2.
  Body bone mass of participants will be analyzed by bioimpedance and reported in kilograms.
The incidence of catarrhal episodes | Clinical Investigation Day 1 and Clinical Investigation Day 2.
  The number of catarrhal episodes will be registrated through a questionnaire designed for that purpose.
The gravity of catarrhal episodes | Clinical Investigation Day 1 and Clinical Investigation Day 2.
  The gravity (mild/half /serious) of catarrhal episodes will be registrated through a questionnaire designed for that purpose.
Gastrointestinal symptoms | Clinical Investigation Day 1 and Clinical Investigation Day 2.
  Gastrointestinal symptoms will be registrated through Gastrointestinal Symptoms Rating Scale questionnaire, which is a questionnaire of 15 items. The questionnaire has a seven-point graded likert-type scale, where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms.
Dietary intake | Clinical Investigation Day 1 and Clinical Investigation Day 2.
  Dietary intake (energy, macronutrients and micronutrients) will be analysed by food frequency questionnaire.
Physical activity | Clinical Investigation Day 1 and Clinical Investigation Day 2.
  Physical activity will be evaluated by the reduced version of the International Physical Activity Questionnaire, which estimates the total physical activity in MET-min/week, time spent sitting and classifies subjects based on their physical activity
Adherence to capsule consumption | Clinical Investigation Day 1 and Clinical Investigation Day 2.
  Adherence will be assessed using the capsule consumption record form.

CONTACTS AND LOCATIONS:
Overall Officials: Fermín Milagro Yoldi, PhD, Principal Investigator — University of Navarra; Idoia Ibero-Baraibar, PhD, Study Chair — University of Navarra; Carlos González-Navarro, Study Chair — University of Navarra; Santiago Navas-Carretero, Study Chair — University of Navarra; Roncesvalles Garayoa, PhD, Study Chair — University of Navarra; Gabriela Arias, Study Chair — University of Navarra; Blanca Martinez, Study Chair — University of Navarra; Salomé Pérez, Study Chair — University of Navarra; María Goñi, Study Chair — University of Navarra
Locations (1):
- Centre for Nutrition Research, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No